CLINICAL TRIAL: NCT03217370
Title: Study on Patient Blood Management in Haematological Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: the pilot study (before the intervention) is completed.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S60580
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Blood Transfusion; Haematology
Keywords: patient blood management; restrictive transfusion

STUDY DESIGN:
Intervention Model Description: observational cross-sectional study with pre and post measurement and in between an interventional phase with education, IT implementations etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all haematologists (Other): There will be only one arm: the haematologists will all be included in the interventional phase.
  Interventions are: 1) rewriting guidelines to order blood components; 2) to show the last hemoglobin value on the orders for erytrocytes and the last platelet count on the orders dor thrombocytes and 3)implementation of a clinical decision support system in the electronic rodering of blood components to stimulate restrictive blood transfusion.
  Interventions: Other: education of guidelines

INTERVENTIONS:
Other: education of guidelines — * Guidelines will be updated and education will be given to haematologists in several ways.
  * ICT implementations: a) last result of haemoglobin and platelet count will be shown on the electronic blood order; b) an electronical clinical decision support system will be implemented to order blood components
  Other Names: ICT implementations in the electronic patient file

SUMMARY:
The investigators noticed a variable prescription of blood components to haematological patients in the hospital. This study will analyze the prescription and administration of blood components to Haematological patients (pre measurement). Based on these results guidelines on transfusion triggers will be updated and educated to the physicians and new ICT (information and communications technology) implementations will be added to the electronic order for blood components. The investigators hope to see afterwards (post measurement) a more stable prescription and administration of blood components and a more economic use of blood components.

DETAILED DESCRIPTION:
This study is set up as a first step of implementing patient blood management (PBM) in this hospital. PBM is an evidence-based, multidisciplinary approach to optimizing the care of patients who might need transfusion. Not only in pre/per/postoperative setting but also in haematology PBM guidelines can be implemented. Examples are: use of a restrictive haemoglobin trigger for red blood cells (RBC) transfusion, single use policy for the administration of RBC and platelets, administration only for correct indications (including the introduction of an electronic clinical decision support system for ordering blood components), ...

ELIGIBILITY:
Inclusion Criteria:

* all adult patients hospitalised at the haematology wards of the University Hospitals of Leuven (UZ Leuven) between 01/08/2017 and 31/07/2018 (pre measurement) and between between 01/08/2019 and 31/07/2020 (post measurement)

Exclusion Criteria:

* ambulatory patients
* patients without blood transfusion administered in their hospitalised period
* patients with no haematological illness that were hospitalised at the haematological wards

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
how do haematologists prescribe blood components? | up to 1 year pre measurement and up to 1 year post measurement
  The investigators use a questionaire (15-20 questions) to evaluate how haematologists prescribe red blood cells and platelets. Do they analyze the haemoglobin and platelet count before and after each blood transfusion? Do they apply single unit policy for RBC and platelet transfusions? Which triggers are used for RBC and platelet transfusion? Which guidelines are followed? The investigators will send this questionnaire to all haematologists (including haematologists in training) in 2017 (premeasurement) and in 2019-2020 (postmeasurement).
  The investigators will also use data (which is already available in the patient files) about blood transfusion to evaluate the ordering and administration of blood components during 1 year. For which indication is blood ordered? Is the Haemoglobin level known before the order is send to the blood bank?

SECONDARY OUTCOMES:
what's the effect of the interventional phase? | up to 1 year (post measurement)
  The investigators will again use data (which is already available in the patient files) about blood transfusion to evaluate the ordering and administration of blood components during 1 year after the intervention phase. For which indication is blood ordered? Is the Haemoglobin level known before the order is send to the blood bank? Did the interventions lead to less prescriptions/administrations of blood components and more single unit transfusion? We will use SPSS for statistical analysis (frequencies, percentages and means, scatter plots)

CONTACTS AND LOCATIONS:
Overall Officials: Els Costermans, MD, Principal Investigator — advanced clinical nurse specialist
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No